CLINICAL TRIAL: NCT02939794
Title: The Effect of Intra Venus Ferric Carboxymaltose Preoperative on Hemoglobin and Blood Transfusion Post Cardiac Surgery
Brief Title: The Effect of Ferric Carboxymaltose on Hemoglobin and Blood Transfusion in Cardiac Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Carmel Medical Center (Other); The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Principal Investigator, Gil Bolotin MD, prof, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105-02
Record Dates: First submitted 2016-05-31; First posted 2016-10-20 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Anemia
Keywords: cardiac surgery; hemoglobin; iron
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ferinject (Active Comparator): -Patients will receive 1000 mg of a ferric carboxymaltose (Ferinject type) intravenously approximately 24 hours prior to surgery
  Interventions: Drug: Ferinject
- placebo (Placebo Comparator): Patients will receive a placebo drug intravenous approximately 24 hours before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferinject — 1000 mg of a ferric carboxymaltose (Ferinject type) intravenously approximately 24 hours prior to surgery
  Other Names: ferric carboxymaltose
  Arms: ferinject
Drug: Placebo — Saline (normal saline, sodium chloride)
  Other Names: Saline
  Arms: placebo

SUMMARY:
Anemia after cardiac surgery is a vast phenomena. More than 70% of the patients who under went surgery represented with hemoglobin less than 8 mg/dl (the cutoff for blood transfusion) and more than 80% of the patients receives at least one unit of red blood cell transfusion.

There were number of attempts to prevent the postoperative anemia by giving erythropoietin, Iron per os and intra venus iron. non of the above have shown increase in Hemoglobin after the cardiac surgery.

DETAILED DESCRIPTION:
Research Objectives

The study objectives are:

1. Determine hemoglobin values in non-anemic patients given ferric Carboxymaltose prior to and post heart surgery.
2. Determine the effect of ferric Carboxymaltose in non-anemic patients prior to surgery on the number of blood units administer postoperation.

Research Methods Prospective, randomized, double-blind, placebo-controlled research. All patients who are in the cardiac surgery department for bypass surgery, valve replacement surgery or combined surgery will be eligible to participate in the study. The study will be presented and explained to all patients and, if they consent, patients will be divided into two random groups. One group will receive Ferinject IV 24-48 hours prior to surgery. The second group will receive a placebo drug in the same time period as when the drug Ferinject is administered.

The Population Studied All patients aged 18 or older hospitalized at the Rambam Medical Center and are candidates for open-heart surgery (coronary artery bypass, valve, combined).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Patient candidates for open heart surgery (coronary artery bypass, valve replacement, or a combination of both).
3. Hemoglobin above 12g/dL in women and above than 13g\dL in men.

Exclusion Criteria:

1. Patients who require emergency heart surgery.
2. Patients who are not hemodynamically stable or intubated pre-operatively.
3. Patients with a known sensitivity to iron.
4. Patients with a known history of allergies (rashes, etc.).
5. Patients with liver failure (alanine aminotransferase> 3 times normal).
6. Patients with cirrhosis.
7. Patients with an active infection.
8. Patients with rheumatoid arthritis and indications of an active infection.
9. Pregnant women.
10. Lactating women.
11. Patients with anemia prior to surgery for any reason (B12 deficiency or folic acid deficiency).
12. Patients participating in another drug trial.
13. Patients treated with iron who took medication within the four weeks prior to surgery.
14. Patients who received a blood transfusion in the four weeks prior to surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
In order to determine the effect of ferric Carboxymaltose in non-anemic patients prior to surgery on the number of blood units administer postoperation, we will count the number of red packed cells and hemoglobin will be measured in gr\dl% | 2 years
  • All patients post heart surgery will be admitted to the intensive care unit cardiac surgery for a minimum of 48 hours. The unit has regular and routine monitoring for blood tests (blood chemistry panel, coagulation) and blood gases.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Friedman T, Dann EJ, Bitton-Worms K, Makhoul M, Glam R, Weis A, Tam DY, Bolotin G. Intravenous iron administration before cardiac surgery reduces red blood cell transfusion in patients without anaemia. Br J Anaesth. 2023 Dec;131(6):981-988. doi: 10.1016/j.bja.2023.09.007. Epub 2023 Oct 12. PMID 37838604